CLINICAL TRIAL: NCT06539546
Title: Shade Matching and Patient Satisfaction of Yttria Stabilized Multilayered Zirconia and Lithium Disilicate Restorations: a Randomized Controlled Clinical Trial
Brief Title: Shade Matching and Patient Satisfaction of Yttria Stabilized Multilayered Zirconia and Lithium Disilicate Restorations
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Yasmin Mohamed, Principal Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PROSF 3.3.6
Record Dates: First submitted 2024-07-29; First posted 2024-08-06 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: Mutilated Teeth; Endodontically Treated Teeth
Keywords: Shade match; patient satisfaction; Yttria stabilized multilayered zirconia; Lithium disilicate
MeSH Terms: conditions — Tooth, Nonvital; Patient Satisfaction

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Yttria stabilized multilayered (YML) zirconia restorations (Experimental): Full coverage Yttria stabilized multilayered (YML) zirconia restorations will be fabricated on a tooth requiring full coverage in the esthetic zone.
  Interventions: Other: Yttria stabilized multilayered (YML) zirconia restorations
- Lithium disilicate restorations (Experimental): Full coverage Lithium disilicate restorations will be fabricated on a tooth requiring full coverage in the esthetic zone.
  Interventions: Other: Lithium disilicate restorations

INTERVENTIONS:
Other: Yttria stabilized multilayered (YML) zirconia restorations — Yttria stabilized multilayered zirconia restorations were claimed to have high strength and esthetics at the same time but no clinical studies were conducted yet to prove its high esthetic properties
  Arms: Yttria stabilized multilayered (YML) zirconia restorations
Other: Lithium disilicate restorations — Lithium disilicate reinforced glass ceramics are considered a gold standard for monolithic esthetic restorations.
  Arms: Lithium disilicate restorations

SUMMARY:
The aim of the study is to determine whether Yttria stabilized multilayered zirconia restorations will differ from lithium disilicate restorations in shade matching and patient satisfaction in patients requiring full coverage restorations.

DETAILED DESCRIPTION:
Steps in short: Single tooth in the esthetic zone requiring full coverage crown is prepared to receive an all-ceramic crown, The restorations will be divided into two groups: I: Teeth receiving restorations fabricated from Lithium disilicate II: Teeth receiving restorations fabricated from yttria stabilized multilayered zirconia. Shade will be measured using intraoral spectrophotometer and evaluated. The colour difference (ΔE) will be calculated for each sample using the following equation: ΔE =[(ΔL) ²+(Δa) ² + (Δb) ²] ½, ΔE (perceptibility threshold) will be evaluated for each group. Participant timeline the patient will be treated in visits designated as follows: Visit 1: Preoperative records, face-to-face adherence reminder session, clinical, radiographic for examination, intraoral photographs and primary impression (Alginate impression) diagnostic cast construction. Visit 2: teeth preparation and secondary impression using addition silicone rubber base material and temporary restoration. Visit 3: placement and permanent cementation of the final restoration using resin cement.

ELIGIBILITY:
Inclusion criteria:

1. Age range of the patients from 20-60 years old; able to read and sign the informed consent document, illiterate patient will be avoided.
2. Patients able physically and psychologically to tolerate conventional restorative procedures.
3. Patients with no active periodontal or pulpal diseases, having teeth with good restorations.
4. Patients with teeth problems indicated for full coverage restoration (coronal fracture where partial coverage would lack retention, malposed or malformed teeth).
5. Patients with root canal treated teeth requiring full coverage restorations.
6. Patients willing to return for follow-up examinations and evaluation.

Exclusion Criteria:

1. Patients in the growth stage with partially erupted teeth.
2. Patients with poor oral hygiene and motivation.
3. Patients with psychiatric problems or unrealistic expectations (patient that has phobia from dental treatments or needle bunch).
4. Patients suffer from parafunctional habits.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 22 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-09-01 (Estimated)

PRIMARY OUTCOMES:
Color difference | immediate after cementation
  By Intraoral Spectrophotometer, color difference between the restoration and the adjacent or contralateral natural tooth will be measured by the unit (ΔE), (ΔE) will be measured for each sample.

SECONDARY OUTCOMES:
Patient satisfaction | immediate after cementation
  By Visual Analogue Scale, with score range from 1 to 10 , where 1 is the worst (lowest satisfaction) and 10 is the best (highest satisfaction).